CLINICAL TRIAL: NCT01963013
Title: A Pilot Study of Non-returning Catheter Valve for Reducing Catheter-associated Urinary Tract Infection in Critically-ill Patients
Brief Title: Non-returning Catheter Valve for Reducing CAUTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Anupol Panitchote, Anupol Panitchote, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAUTI-001
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Catheter Associated Urinary Tract Infection; Critically Ill Patients
Keywords: Non-returning catheter valve; Catheter associated urinary tract infection; Critically ill patients; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-returning catheter valve (Experimental): Non-returning catheter valve (UnometerTM SafetiTM Plus) was used in experimental group only.
  Interventions: Device: Non-returning catheter valve
- Conventional urine bag (Active Comparator): Conventional urine bag hasn't the non-returning catheter valve.
  Interventions: Device: Conventional urine bag

INTERVENTIONS:
Device: Non-returning catheter valve
  Other Names: UnometerTM SafetiTM Plus
  Arms: Non-returning catheter valve
Device: Conventional urine bag
  Arms: Conventional urine bag

SUMMARY:
This study was to determine efficacy of the non-returning catheter valve for reducing catheter associated urinary tract infection compared with conventional urine bag in critically ill patients.

DETAILED DESCRIPTION:
Non-returning catheter valve (generic name) used UnometerTM SafetiTM Plus (trade name)

ELIGIBILITY:
Inclusion Criteria:

* The participants who age more than 18 year and admitted to the medical intensive care unit or intermediate care unit
* All participants must be retained the urinary catheter.

Exclusion Criteria:

* The participants were diagnosed urinary tract infection before retention of the urinary catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence density of the catheter associated urinary tract infection (CAUTI) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Srinagarind hospital, Muang, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Panitchote A, Charoensri S, Chetchotisakd P, Hurst C. Pilot study of a non-return catheter valve for reducing catheter-associated urinary tract infections in critically ill patients. J Med Assoc Thai. 2015 Feb;98(2):150-5. PMID 25842795